CLINICAL TRIAL: NCT01063543
Title: Population Pharmacokinetics of Fondaparinux Administered at Prophylactic Doses After Major Orthopedic Surgery in Everyday Practice
Brief Title: Pharmacokinetics of Fondaparinux in Patients With Major Orthopedic Surgery
Acronym: POP-A-RIX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Pr Patrick MISMETTI, Centre Hospitalier Universitaire de Saint Etienne
Other Study IDs: 0601069
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Orthopedic Surgery
Keywords: fondaparinux; orthopedic surgery; patients with major orthopedic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for anti-Xaactivity measure
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with blood sample: Patients with major orthopedic surgery and prophylactic doses of fondaparinux who have 3 blood sample during their hospitalization to measure anti-Xa activity

SUMMARY:
Fondaparinux is a synthetic antithrombotic agent with specific anti-factor Xa activity. A population pharmacokinetic model of fondaparinux, based on data obtained in patients included in phase II/III trials, has been described. However, the validity of this model in everyday practice needed to be confirmed. This study was a multicenter, prospective cohort study in consecutive orthopedic patients treated with 2.5 mg of fondaparinux. Anti-Xa activities were recorded in 809 patients. Population parameters and inter-individual variability were estimated using NONMEM VI software. A two-compartment model with first-order absorption best described fondaparinux pharmacokinetics. Covariates partly explaining inter-individual variability were body weight, age and creatinine clearance estimated by the simplified Modification of Diet in Renal Disease formula. A body weight less than 50 kg and moderate renal failure increased drug exposure. These results suggest that fondaparinux pharmacokinetics need to be confirmed in patient populations not fully assessed in phase II/III studies

ELIGIBILITY:
Inclusion Criteria:

* patient who need leg major orthopedic surgery
* age > 18 years
* patient who need prophylactic doses of fondaparinux

Exclusion Criteria:

* contra-indication to fondaparinux
* renal insufficiency

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with major orthopedic surgery who need prophylactic doses of fondaprinux
Sampling Method: Non-Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2004-09; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To determine an anti-Xa activity value which is predicted of a haemorrhage risk | day 9

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, Pr, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - CHARRET Françoise, Annonay
  - PEGOIX Michel, Caen
  - ROSENCHER Nadia, Paris
  - PETIT Pierre-Yves, Pierre-Bénite
  - BARRE Jeanne, Reims
  - MAITRE Anne-Marie, Rouen
  - BAYLOT Denis, Saint-Etienne
  - ZUFFEREY Paul, Saint-Etienne